CLINICAL TRIAL: NCT04057339
Title: Influence of Time-restricted Eating (TRE) on Circadian Regulation of Glucose Homeostasis and Mitochondrial Function - The TIMET Study
Brief Title: The Influence of Time-Restricted Eating in Patients With Metabolic Syndrome
Acronym: TIMET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Salk Institute for Biological Studies (Other)
Responsible Party: Principal Investigator, Pam Taub, MD, Associate Professor of Medicine, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 181088; 1R01DK118278-01 (NIH)
Record Dates: First submitted 2019-04-02; First posted 2019-08-15 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Metabolic Syndrome; Pre-Diabetes
Keywords: Time Restricted Eating; Circadian Rhythm; Glucose Homeostasis; Mitochondrial Function; Fasting
MeSH Terms: conditions — Metabolic Syndrome; Glucose Intolerance; Intermittent Fasting; Fasting | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SOC (Standard of Care) (Placebo Comparator): Everyone in this arm will receive standard of care nutritional behavioral counseling and will be required to log their caloric intake through the use of a smartphone app.
  Interventions: Behavioral: Standard of Care
- TRE + SOC (Experimental): Everyone in this arm will receive standard of care nutritional behavioral counseling and will implement a daily 8-10-hour window within which they must consume their calories. They will also be required to log their caloric intake through the use of a smartphone app.
  Interventions: Behavioral: Time Restricted Eating + Standard of Care

INTERVENTIONS:
Behavioral: Time Restricted Eating + Standard of Care — Participants in this arm will adhere to a daily, consistent 8-10-hr eating window for the course of the study as well as receive nutritional counseling from the study dietitian.
  Other Names: Time Restricted Eating
  Arms: TRE + SOC
Behavioral: Standard of Care — Participants in this arm will receive nutritional counseling from the study dietician, but will not be required to adopt a 8-10-hr eating window.
  Arms: SOC (Standard of Care)

SUMMARY:
In a randomized controlled trial, the investigators intend to measure the health impact of TRE in patients with metabolic syndrome (with three or more of the following criteria: increased waist circumference, abnormal cholesterol levels, elevated blood pressure, or elevated blood sugar), who habitually eat for more than 14 hours every day. Patients will be randomly assigned to a control group of behavioral nutrition counseling (standard of care) or the intervention group of behavioral nutrition counseling with the addition of adopting a 8-10 hour eating window for 12 weeks (TRE).

DETAILED DESCRIPTION:
Circadian rhythms optimize nutrient homeostasis by orchestrating catabolic and anabolic metabolism to appropriate times of the 24 hour day. Chronic circadian rhythm disruption predisposes individuals to metabolic diseases including obesity and type 2 diabetes. Conversely, maintaining a daily rhythm of feeding and fasting cycles sustains a robust circadian rhythm which improves cellular bioenergetics and results in improved metabolism. Time-restricted eating (TRE) is a specific feeding-fasting pattern in which feeding is restricted to 8-12 hours a day.

At the beginning and end of the study (which will be three months in duration), the following parameters will be measured: height, weight, body mass index, percent body fat, waist/hip circumference and blood pressure. Blood sugar levels will be monitored continuously for 2 weeks at a time at the beginning and end of the study using a continuous glucose monitor. Additionally, a dual energy X-ray absorptiometry (DXA) scan will be used to collect information about body composition. Information will be collected about the mitochondria with a muscle biopsy. Participants will use a smartphone application (called myCircadianClock (mCC), developed by the Salk Institute) to keep track of food/beverage intake and will wear a wrist-worn actigraphy device to monitor physical activity levels and sleep.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years
2. 41 ≥ BMI ≥ 25 AND
3. Metabolic syndrome, as defined as presence of 3 or more of the following criteria:

   Elevated fasting plasma glucose ≥ 100 mg/dL and/or HbA1c ≥ 5.7% < 7.1% Elevated waist circumference: In Asians: ≥ 90 cm in men, ≥ 80 cm in women, all other races: ≥ 102 cm in men, ≥ 88 cm in women Fasting plasma triglycerides ≥ 150 mg/dL, or on drug treatment for elevated triglycerides Reduced High-density lipoprotein (HDL)-cholesterol < 40 mg/dL in males or < 50 mg/dL in females, or drug treatment for reduced HDL-cholesterol Elevated blood pressure, Systolic blood pressure ≥ 135 mm Hg and/or diastolic blood pressure ≥ 85 mm Hg or drug treatment for hypertension
4. Own a smartphone (Apple iOS or Android OS)
5. Baseline eating period ≥ 12 hour window
6. If patients are on cardiovascular medications (HMG CoA reductase inhibitors (statins), other lipid modifying drugs (including over the counter drugs such as red yeast rice and fish oil), anti-hypertensive, anti-diabetes drugs), no dose adjustments will be allowed during the study period.

Exclusion Criteria:

1. Taking insulin within the last 6 months.
2. Manifest diabetes, defined as HbA1c > 7.0% given a 0.3% margin of error in lab readings, or diagnosis of diabetes.
3. Known inflammatory and/or rheumatologic disease.
4. Active tobacco abuse or illicit drug use or history of treatment for alcohol abuse.
5. Pregnant or breast-feeding women.
6. Shift workers with variable (e.g. nocturnal) hours.
7. Caregivers for dependent requiring frequent nocturnal care/sleep interruptions.
8. Planned travel to a time zone with greater than a 3-hour difference during study period.
9. History of major adverse cardiovascular event within the past 1 year (acute coronary syndrome (ACS), percutaneous coronary intervention, coronary artery bypass graft surgery, hospitalization for congestive heart failure, stroke/transient ischemic attack (TIA)).
10. Uncontrolled arrhythmia (i.e. rate-controlled atrial fibrillation/atrial flutter are not exclusion criteria).
11. History of thyroid disease requiring dose titration of thyroid replacement medication(s) within the past 3 months (i.e. hypothyroidism on a stable dose of thyroid replacement therapy is not an exclusion).
12. History of adrenal disease.
13. History of malignancy undergoing active treatment, except non-melanoma skin cancer.
14. Known history of type I diabetes.
15. History of eating disorder(s).
16. History of cirrhosis.
17. History of stage 4 or 5 chronic kidney disease or requiring dialysis.
18. History of HIV/AIDS.
19. Currently enrolled in a weight-loss or weight-management program.
20. On a special or prescribed diet for other reasons (e.g. Celiac disease).
21. Currently taking any medication that is meant for, or has known effect on, appetite.
22. Any history of surgical intervention for weight management.
23. Uncontrolled psychiatric disorder (including history of hospitalization for psychiatric illness).
24. A score of >16 on the Epworth Sleepiness Scale (ESS).
25. Depression determined by the Beck Depression Inventory (BDI) (unless previously diagnosed and well-controlled).
26. Failure to use the smartphone app for documentation (defined as <2 meals/day for ≥3 days during baseline).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Change in glucose levels assessed via HbA1c | Baseline and 14 weeks
  HbA1c (%)
Change in glycemic parameters | Baseline and 14 weeks
  Glycemic parameters assessed via fasting glucose (mg/dL), HOMA-IR, Insulin (mIU/L), and continuous glucose monitors (CGM).

SECONDARY OUTCOMES:
Change in LDL particle number | Baseline and 14 weeks
  LDL particle number (nmol/L) via NMR lipoprofile
Change in LDL cholesterol | Baseline and 14 weeks
  LDL cholesterol (mg/dl)
Change in HDL cholesterol | Baseline and 14 weeks
  HDL cholesterol (mg/dl)
Change in Triglycerides | Baseline and 14 weeks
  Triglycerides (mg/dl)
Change in body composition by DXA | Baseline and 14 weeks
  Lower abdominal fat mass as assessed by dual-energy X-ray absorptiometry (DXA).
Change in hs-CRP | Baseline and 14 weeks
  High sensitivity C-reactive protein (mg/L)

OTHER OUTCOMES:
Change in mitochondrial structure and gene expression in skeletal muscle | Baseline and 14 weeks
  Mitochondrial structure and gene expression in skeletal muscle as assessed by skeletal muscle biopsies.

CONTACTS AND LOCATIONS:
Overall Officials: Pam Taub, MD, Principal Investigator — Associate Professor of Medicine
Locations (1):
- Altman Clinical and Translational Research Institute, La Jolla, California, United States

REFERENCES:
- [Derived] Manoogian ENC, Wilkinson MJ, O'Neal M, Laing K, Nguyen J, Van D, Rosander A, Pazargadi A, Gutierrez NR, Fleischer JG, Golshan S, Panda S, Taub PR. Time-Restricted Eating in Adults With Metabolic Syndrome : A Randomized Controlled Trial. Ann Intern Med. 2024 Nov;177(11):1462-1470. doi: 10.7326/M24-0859. Epub 2024 Oct 1. PMID 39348690
- [Derived] Taub PR, Panda S. Time for better time-restricted eating trials to lessen the burden of metabolic diseases. Cell Rep Med. 2022 Jun 21;3(6):100665. doi: 10.1016/j.xcrm.2022.100665. PMID 35732151

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2021-12-02): https://cdn.clinicaltrials.gov/large-docs/39/NCT04057339/Prot_ICF_000.pdf